CLINICAL TRIAL: NCT03751059
Title: An Investigator-Initiated Multicenter Prospective Clinical Trial to Examine the Efficacy of Peri-operative NSAID vs Steroid Treatment in Trabeculectomy Wound Management
Brief Title: NSAID vs Steroid in Trabeculectomy Wound Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cindy Hutnik (Other)
Collaborators: Glaucoma Research Society of Canada (Other)
Responsible Party: Sponsor-Investigator, Cindy Hutnik, Principal Investigator, Ivey Eye Institute
Organization: Ivey Eye Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TWM
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — bromfenac; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAID (Active Comparator): Bromfenac 0.07% Oph Susp: used from one week post-op to three months post-op
  Interventions: Drug: Bromfenac 0.07% Oph Susp
- Steroid (Active Comparator): Dexamethasone: used from one week post-op to three months post-op
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Bromfenac 0.07% Oph Susp — Bromfenac 0.07% Oph Susp to be used post-operatively (week 1 to month 3) by one treatment group.
  Other Names: Bromfenac
  Arms: NSAID
Drug: Dexamethasone — Topical dexamethasone to be used by all study participants for one week pre-trabeculectomy and by all study participants for one week post-trabeculectomy. At one week post-op, one of the treatment groups will continue to dose with dexamethasone.
  Arms: Steroid

SUMMARY:
This study will examine the efficacy of steroid vs NSAID treatment in relation to trabeculectomy wound management. Eligible study participants will be randomized to receive either steroid or NSAID topical treatment one week post-trabeculectomy. Each group will dose with their assigned study treatment until three months post-trabeculectomy. Study participants will be followed for twelve months post-trabeculectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 years
* Uncontrolled open angle glaucoma
* Scheduled to undergo stand-alone trabeculectomy
* No previous incisional glaucoma surgery
* No ocular surgery of any kind in prior 6 months

Exclusion Criteria:

* steroids and/or NSAIDs contraindicated
* poor corneal epithelial health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Target IOP | 12 months
  the proportion of patients achieving a target IOP range (≤21, ≤18, ≤15 or ≤12 mmHg) at 12 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Hutnik, MD, Principal Investigator — Ivey Eye Institute